CLINICAL TRIAL: NCT03856840
Title: Evaluation of Cytokines and Immunoglobulins in Serum and Blister Fluids Appeared Before Treatment and Subsequently Under Treatment in Bullous Pemphigoid
Brief Title: Cytokines in Blister Fluids of Bullous Pemphigoid (BP)
Acronym: BP
Status: Completed | Type: Observational
Sponsor: Mahmut Can Koska (Other)
Responsible Party: Sponsor-Investigator, Mahmut Can Koska, Assistant Doctor, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Other Study IDs: 2018/0181
Record Dates: First submitted 2019-02-19; First posted 2019-02-27 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Pemphigoid, Bullous
Keywords: Pemphigoid, Bullous; Bullous Pemphigoid; Blister Fluid; Eosinophil Cationic Protein; Tumor Necrosis Factor-alpha; Anti-BP180; Disease activity; Disease severity
MeSH Terms: conditions — Pemphigoid, Bullous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Blister Fluid: Blister fluids will be obtained from all enrolled patients in specific three intervals: Before treatment, 4-7. and 8-14. days of treatment in 24 hours after they appear.
  Bullae of only one individual day will be selected for each interval to study if they appeared.
  Blood Serum: Blood serum will be obtained from all enrolled patients before treatment, seventh day of treatment and fourteen day of treatment.
  Obtaining blood serum from patients was added to study afterward. New ethical committee approval was received for that modification in recruitment status at May 17, 2018. Thus blood serum weren't obtained patients who were recruited before that approval. But other specimens obtained from these patients will be included study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bullous Pemphigoid Patients: Bullae and blood serum, which are obtained before and under treatment, will be compared in each other regardless of any condition.

SUMMARY:
This study investigates the differences of Eosinophil Cationic Protein, Tumor Necrosis Factor-alpha and Anti-BP180-NC16A IgG levels of blister fluids in Bullous Pemphigoid patients which appeared before and under treatment subsequently. These molecules will also be measured in blood serum before and under treatment. Changes of titers in serum and differences between blister fluids will be compared to observe whether correlation exists between them. These measures will also be compared between groups of responders and non-responders to the first-line treatment options to analyze correlation with treatment success.

DETAILED DESCRIPTION:
Bullous Pemphigoid is an auto-immune bullous disorder in which auto-antibodies to hemidesmosomes, complement pathway, inflammatory cells and mediators play a crucial roles for disease pathogenesis.

Anti-BP180-NC16A IgG is an antibody that it primarily triggers inflammatory reactions and complement cascade in bullae development and plays major roles in disease pathogenesis. It is secreted by plasma cells which is induced by T-helper 2 cells and their cytokines in serum and lesional tissue. Anti-BP180 antibody detection in serum is very important in diagnosis and titers correlate with disease activity. Anti-BP180 antibody can also be detected in blister fluids and it may aid diagnosis.

Eosinophil cationic Protein is a cytokine and secreted by Eosinophil which is found in abundant numbers and correlated with tissue damage in Bullous Pemphigoid lesions. Serum titers of Eosinophil Cationic Protein has a correlation with disease activity and it is higher in blister fluid than serum. Tumor Necrosis Factor-alpha is an another cytokine which is secreted from inflammatory cells initially after inflammatory cascade is triggered. It is also found increased in serum blister fluids. Tumor necrosis factor-alpha is associated with clinical severity in bullous pemphigoid.

In Bullous Pemphigoid, development of bulla is required to be stopped if treatment will be considered as successful. Nevertheless smaller, more rapidly healing vesicles and bullae appear under treatment which are not regarded as findings of treatment failure. In this study we will measure Eosinophil Cationic Protein, Tumor Necrosis Factor-alpha and Anti-BP180-NC16A IgG levels with E.L.I.S.A. technique in these subsequently appeared blisters if they will appear and compare them with pretreatment blisters. We will also measure levels of these molecules in blood serum before and under treatment. We will analyze corralation between blood serum and blister fluids. Also we will compare responder patients and non-responder patients to first-line treatment options to observe correlation of changes and differences in these body fluids with treatment success.

ELIGIBILITY:
Inclusion Criteria:

* All patiens presented to clinics who is diagnosed with Bullous Pemphigoid by findings of clinical, histopathological, Direct Immunoflorescent evaluation.
* All relapsed/flared Bullous Pemphigoid patients.
* Patients who accept the terms and conditions and sign consent form.

Exclusion Criteria:

* Patients who are received treatment before presenting clinics where the study is conducted.
* Patients who reject to join to study and the terms and condition
* Patients who leave the study by own decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Bullous Pemphigoid patients presented to concerning clinics who accept the terms and definitions and sign consent form.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-08-27 (Actual)

PRIMARY OUTCOMES:
Titers of Eosinophil Cationic Protein in blister fluid and blood serum | 14 Days
  Calculated of measurements of Eosinophil Cationic Protein (pg/ml) by ELISA technique in blister fluids and serums that obtained before treatment and under first and second weeks of treatment.
Titers of Tumor Necrosis Factor-alpha in blister fluid and blood serum | 14 Days
  Calculated of measurements of Tumor Necrosis Factor-alpha (pg/ml) by ELISA technique in blister fluids and serums that obtained before treatment and under first and second weeks of treatment.
Titers of Anti-BP180-NC18A IgG in blister fluid and blood serum | 14 Days
  Calculated of measurements of Anti-BP180-NC18A IgG (U/ml) by ELISA technique in blister fluids and serums that obtained before treatment and under first and second weeks of treatment.

SECONDARY OUTCOMES:
Time to control of disease activity | Up to 4 weeks
  Time interval between initiation of treatment and control of disease activity/beginning of consolidation phase
Consolidation phase of Outcome Measures for Bullous Pemphigoid | 14 days
  Time interval between control of disease activity and end of consolidation phase.
Treatment Failure | 4 week
  Development of nontransient lesions that heal in more than one week, continued extension of old lesions, failure of established lesions to begin to heal or continued pruritus despite of Treatment of one month.
Relapse/Flare | Up to one year
  Appearance of more than three lesions per month or at least one large eczematous lesion or urticarial plaques that do not heal within one week, or extension of established lesions or daily pruritus in patient who was achieved disease control
Bullous Pemphigoid disease severity assessment | One day
  This assessment will depend on multiple factors according to more than one classification. Patients will be separated to mild, moderate, severe conditions according to their clinical findings.
  Mild: Involvement of less than %10 of skin surface area and appearance of less than 10 bullae in each day. Both feature will be necessary to regard individual patient's disease as mild.
  Moderate: Involvement of %10-30 of skin surface area and appearance of less than 10 bullae in each day. Both feature will be necessary to regard individual patient's disease as moderate.
  Severe: Involvement of more than %30 of skin surface area or appearance of more than 10 bullae in each day or B.P.D.A.I. score more than 56 (without Visual analogue score of pruritus). Existence of even one of this findings will ve sufficient to regard individual patient's disease as severe.
Bullous Pemphigoid Disease Area Index (B.P.D.A.I.) | Up to one year
  BPDAI is an index to assess disease area and severity depending on involvement of mucosa and skin region, lesion number and size. Minimum score is 0 and maximum score is 360.
  This index will be calculated at before treatment, second week and fourth week of treatment. After first month it will be calculated in each follow-up visit.
Bullous Pemphigoid Disease Area Index (B.P.D.A.I.)-Damage score | Up to one year
  Scars of previous lesions are also included to this index, minimum score is 0 and maximum score is 12.
  This index will be calculated at before treatment, second week and fourth week of treatment. After first month it will be calculated in each follow-up visit.
Bullous Pemphigoid Disease Area Index (B.P.D.A.I.)-Pruritus score | Up to one year
  Visual analogue score of pruritus is also part of this index. Minimum score is 0 and maximum score is 10. This score will be assessed for last 24 hours, last one week, last one month one by one; thus maximum score will be 30.
  This index will be calculated at before treatment, second week and fourth week of treatment. After first month it will be calculated in each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Salih Gurel, Professor, Study Director — Istanbul Medeniyet University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medeniyet University Goztepe Training and Research Hospital, Istanbul, Kadikoy
  - Istanbul Training and Research Hospital, Istanbul, Samatya

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bernard P, Antonicelli F. Bullous Pemphigoid: A Review of its Diagnosis, Associations and Treatment. Am J Clin Dermatol. 2017 Aug;18(4):513-528. doi: 10.1007/s40257-017-0264-2. PMID 28247089
- [Background] Bagci IS, Horvath ON, Ruzicka T, Sardy M. Bullous pemphigoid. Autoimmun Rev. 2017 May;16(5):445-455. doi: 10.1016/j.autrev.2017.03.010. Epub 2017 Mar 8. PMID 28286109
- [Background] Schmidt E, Zillikens D. Pemphigoid diseases. Lancet. 2013 Jan 26;381(9863):320-32. doi: 10.1016/S0140-6736(12)61140-4. Epub 2012 Dec 11. PMID 23237497
- [Background] Schmidt E, della Torre R, Borradori L. Clinical features and practical diagnosis of bullous pemphigoid. Dermatol Clin. 2011 Jul;29(3):427-38, viii-ix. doi: 10.1016/j.det.2011.03.010. PMID 21605808
- [Background] Marzano AV, Tedeschi A, Fanoni D, Bonanni E, Venegoni L, Berti E, Cugno M. Activation of blood coagulation in bullous pemphigoid: role of eosinophils, and local and systemic implications. Br J Dermatol. 2009 Feb;160(2):266-72. doi: 10.1111/j.1365-2133.2008.08880.x. Epub 2008 Oct 20. PMID 18945300
- [Background] Engineer L, Bhol K, Kumari S, Razzaque Ahmed A. Bullous pemphigoid: interaction of interleukin 5, anti-basement membrane zone antibodies and eosinophils. A preliminary observation. Cytokine. 2001 Jan 7;13(1):32-38. doi: 10.1006/cyto.2000.0791. PMID 11145840
- [Background] Provost TT, Tomasi TB Jr. Immunopathology of bullous pemphigoid. Basement membrane deposition of IgE, alternate pathway components and fibrin. Clin Exp Immunol. 1974 Oct;18(2):193-200. PMID 4619597
- [Background] D'Auria L, Pimpinelli F, Ferraro C, D'Ambrogio G, Giacalone B, Bellocci M, Ameglio F. Relationship between theoretical molecular weight and blister fluid/serum ratio of cytokines and five other molecules evaluated in patients with bullous pemphigoid. J Biol Regul Homeost Agents. 1998 Jul-Sep;12(3):76-80. PMID 9795835
- [Background] Giusti D, Gatouillat G, Le Jan S, Plee J, Bernard P, Antonicelli F, Pham BN. Eosinophil Cationic Protein (ECP), a predictive marker of bullous pemphigoid severity and outcome. Sci Rep. 2017 Jul 6;7(1):4833. doi: 10.1038/s41598-017-04687-5. PMID 28684769
- [Background] Tedeschi A, Marzano AV, Lorini M, Balice Y, Cugno M. Eosinophil cationic protein levels parallel coagulation activation in the blister fluid of patients with bullous pemphigoid. J Eur Acad Dermatol Venereol. 2015 Apr;29(4):813-7. doi: 10.1111/jdv.12464. Epub 2014 Mar 20. PMID 24650303
- [Background] D'Auria L, Pietravalle M, Mastroianni A, Ferraro C, Mussi A, Bonifati C, Giacalone B, Ameglio F. IL-5 levels in the serum and blister fluid of patients with bullous pemphigoid: correlations with eosinophil cationic protein, RANTES, IgE and disease severity. Arch Dermatol Res. 1998 Jan-Feb;290(1-2):25-7. doi: 10.1007/s004030050272. No abstract available. PMID 9522998
- [Background] Dierksmeier U, Frosch PJ, Czarnetzki BM. Eosinophil chemotactic factor (ECF) in blister fluid of dermatological diseases. Br J Dermatol. 1980 Jan;102(1):43-8. doi: 10.1111/j.1365-2133.1980.tb05670.x. PMID 6990957
- [Background] Ameglio F, D'Auria L, Cordiali-Fei P, Mussi A, Valenzano L, D'Agosto G, Ferraro C, Bonifati C, Giacalone B. Bullous pemphigoid and pemphigus vulgaris: correlated behaviour of serum VEGF, sE-selectin and TNF-alpha levels. J Biol Regul Homeost Agents. 1997 Oct-Dec;11(4):148-53. PMID 9582615
- [Background] Murrell DF, Daniel BS, Joly P, Borradori L, Amagai M, Hashimoto T, Caux F, Marinovic B, Sinha AA, Hertl M, Bernard P, Sirois D, Cianchini G, Fairley JA, Jonkman MF, Pandya AG, Rubenstein D, Zillikens D, Payne AS, Woodley D, Zambruno G, Aoki V, Pincelli C, Diaz L, Hall RP, Meurer M, Mascaro JM Jr, Schmidt E, Shimizu H, Zone J, Swerlick R, Mimouni D, Culton D, Lipozencic J, Bince B, Grando SA, Bystryn JC, Werth VP. Definitions and outcome measures for bullous pemphigoid: recommendations by an international panel of experts. J Am Acad Dermatol. 2012 Mar;66(3):479-85. doi: 10.1016/j.jaad.2011.06.032. Epub 2011 Nov 5. PMID 22056920
- [Background] Eming R, Sticherling M, Hofmann SC, Hunzelmann N, Kern JS, Kramer H, Pfeiffer C, Schuster V, Zillikens D, Goebeler M, Hertl M, Nast A, Orzechowski HD, Sardy M, Schmidt E, Sitaru C, Sporbeck B, Worm M. S2k guidelines for the treatment of pemphigus vulgaris/foliaceus and bullous pemphigoid. J Dtsch Dermatol Ges. 2015 Aug;13(8):833-44. doi: 10.1111/ddg.12606. No abstract available. PMID 26213827
- [Background] Zhao CY, Murrell DF. Advances in understanding and managing bullous pemphigoid. F1000Res. 2015 Nov 20;4:F1000 Faculty Rev-1313. doi: 10.12688/f1000research.6896.1. eCollection 2015. PMID 26918143
- [Background] Levy-Sitbon C, Barbe C, Plee J, Goeldel AL, Antonicelli F, Reguiai Z, Jolly D, Grange F, Bernard P. Assessment of bullous pemphigoid disease area index during treatment: a prospective study of 30 patients. Dermatology. 2014;229(2):116-22. doi: 10.1159/000362717. Epub 2014 Jul 5. PMID 25011586
- [Background] Joly P, Roujeau JC, Benichou J, Delaporte E, D'Incan M, Dreno B, Bedane C, Sparsa A, Gorin I, Picard C, Tancrede-Bohin E, Sassolas B, Lok C, Guillaume JC, Doutre MS, Richard MA, Caux F, Prost C, Plantin P, Chosidow O, Pauwels C, Maillard H, Saiag P, Descamps V, Chevrant-Breton J, Dereure O, Hellot MF, Esteve E, Bernard P. A comparison of two regimens of topical corticosteroids in the treatment of patients with bullous pemphigoid: a multicenter randomized study. J Invest Dermatol. 2009 Jul;129(7):1681-7. doi: 10.1038/jid.2008.412. Epub 2009 Jan 29. PMID 19177141
- [Background] Feliciani C, Joly P, Jonkman MF, Zambruno G, Zillikens D, Ioannides D, Kowalewski C, Jedlickova H, Karpati S, Marinovic B, Mimouni D, Uzun S, Yayli S, Hertl M, Borradori L. Management of bullous pemphigoid: the European Dermatology Forum consensus in collaboration with the European Academy of Dermatology and Venereology. Br J Dermatol. 2015 Apr;172(4):867-77. doi: 10.1111/bjd.13717. PMID 25827742